CLINICAL TRIAL: NCT07097246
Title: A Study on the Correlation of Drug Metabolism and Human Body Composition Based on the Bioequivalence Trial of Progesterone Sustained-release Vaginal Gel
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2025-03-223
Record Dates: First submitted 2025-07-17; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observation group

INTERVENTIONS:
Other:  — We do not intervene with the subjects; we only observe their body composition data.

SUMMARY:
The aim of this observational study is to investigate the impact of body composition on the absorption, distribution, and metabolism of drugs. The primary question it seeks to answer is: Does body composition affect the absorption, distribution, and metabolism of drugs? Healthy adult postmenopausal female subjects participating in the quality and efficacy consistency evaluation project for the generic progesterone vaginal sustained-release gel conducted at our hospital will undergo body composition analysis. By combining pharmacokinetic parameters and adverse drug reactions, the study will analyze differences in the metabolism of progesterone vaginal sustained-release gel under various body composition conditions.

During the Phase I clinical trial, under the guidance of the researchers, subjects will use the non-invasive InBody S10 body composition analyzer to obtain body composition data, including but not limited to inorganic salts, muscle mass, lean body mass, body weight, and body fat percentage.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have been successfully enrolled in the bioequivalence trials of Progesterone Sustained-release vaginal gel；
2. Have signed the informed consent form, have a full understanding of the content, process, and risks of this study, and can communicate well with the researchers.

Exclusion Criteria:1:

1）Participants who may not be able to complete the study for other reasons or are deemed by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population consists of subjects who participate in the bioequivalence trial of progesterone vaginal sustained-release gel conducted in the Phase I clinical trial ward of our hospital and who meet the inclusion and exclusion criteria of this trial.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Fat percentage (%) | The day before using drug，and 1 to 4 days after using drug
  Using a body composition analyzer：Inbody S10, non-invasively obtain the subject's body composition data。This instrument applies a very small electrical current to the body and obtains data on various body components based on the characteristics of different body compositions, including fat percentage (%)
Weight | The day before using drug，and 1 to 4 days after using drug
  Weight (kilogram) measured using a body weight scale.
Waist circumference | The day before using drug，and 1 to 4 days after using drug
  Using a body composition analyzer：Inbody S10, non-invasively obtain the subject's body composition data。This instrument applies a very small electrical current to the body and obtains data on various body components based on the characteristics of different body compositions, including Waist circumference（centimeter）

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital and Yuying Children's Hospital Affiliated to Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.